CLINICAL TRIAL: NCT05533931
Title: Comparison of Resistive Breathing Versus Inspiratory Hold Technique in Patients With Chronic Bronchitis
Brief Title: Resistive Breathing Versus Inspiratory Hold Technique in Patients With Chronic Bronchitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahB Muhammad Makhdoom
Record Dates: First submitted 2022-07-14; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Chronic Bronchitis
Keywords: lung infection; resistive breathing; inspiratory hold technique
MeSH Terms: conditions — Bronchitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistive Breathing Training group (Experimental): The patients performed two sessions each of 15 minutes session of resistive breathing for four days a week for six weeks using an inspiratory resistive device. Ask patient to take long slow inspirations while breathing through the resistive device
  Interventions: Other: Resistive Breathing Training group
- inspiratory hold technique (Active Comparator): With the patient in a comfortable position such as side lying or reclined, the therapist may assist the patient by placing both hands on abdominal area to provide proprioceptive feedback. Then in a relaxed tone of voice therapist instructs the patient to sniff quickly through the nose three times with slow, relaxed exhalations
  Interventions: Other: inspiratory hold technique

INTERVENTIONS:
Other: Resistive Breathing Training group — The patients performed two sessions each of 15 minutes session of resistive breathing for four days a week for six weeks using an inspiratory resistive device. Ask patient to take long slow inspirations while breathing through the resistive device
  Arms: Resistive Breathing Training group
Other: inspiratory hold technique — With the patient in a comfortable position such as side lying or reclined, the therapist may assist the patient by placing both hands on abdominal area to provide proprioceptive feedback. Then in a relaxed tone of voice therapist instructs the patient to sniff quickly through the nose three times with slow, relaxed exhalations
  Arms: inspiratory hold technique

SUMMARY:
The aim of the study is to determine the importance and impact of resistive breathing techniques versus inspiratory hold techniques in patients with chronic bronchitis and specially to find out if there are any changes seen in results measured via the incentive spirometer.

DETAILED DESCRIPTION:
Chronic Bronchitis (CB) is defined as a chronic cough and sputum production for at least 3 months a year for 2 consecutive years. It is covered under the umbrella term of Chronic Obstructive Pulmonary Disease (COPD). Chronic bronchitis is thought to be caused by overproduction and hypersecretion of mucus by goblet cells. Epithelial cells lining the airway response to toxic, infectious stimuli by releasing inflammatory mediators and e.g. pro-inflammatory cytokines. During an acute exacerbation of chronic bronchitis, the bronchial mucous membrane becomes hyperemic and edematous with diminished bronchial mucociliary function. This, in turn, leads to airflow impediment because of

luminal obstruction to small airways. The airways become clogged by debris and this further increases the irritation. The characteristic cough of bronchitis is caused by the copious secretion of mucus in chronic bronchitis. Pseudostratified epithelium, highlighting the pseudostratified epithelial cells, goblets cells (shown in blue), then underlying connective tissue.(3) To determine the importance and impact of resistive breathing techniques versus inspiratory hold techniques in patients with chronic bronchitis and specially to find out if there are any changes seen in results measured via incentive spirometer. There are few studies done over it whereas purpose of this research work is to compare these techniques to get better results.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed with chronic bronchitis

  * Clinically stable patients.
  * Both genders.
  * Age 45 to 60 years.
  * Pink puffers included in this study
  * Clients that are involved in research are not allowed for other interventional therapies. They can take their regular medications.
  * Patients diagnosed at least 2 years ago with bronchitis.

Exclusion Criteria:

* • Presence of any genetic disorders (cystic fibrosis).

  * Recent spinal / chest surgery
  * Cardiac issues
  * Fractures of vertebra caused by osteoporosis.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
oxygen saturation | Changes will be assessed at baseline, 3rd week and 6th weeks measured
  amount of oxygen traveling through your body with your red blood cells. Changes will be assessed at baseline, 3rd week and 6th weeks measured
Forced expiratory volume in one second | Changes will be assessed at baseline, 3rd week and 6th weeks measured
  amount of air expired in first one second. Changes will be assessed at baseline, 3rd week and 6th weeks measured
Forced vital capacity | Changes will be assessed at baseline, 3rd week and 6th weeks measured
  the total amount of air exhaled during the FEV test. Changes will be assessed at baseline, 3rd week and 6th weeks measured
FEV1/FVC ratio | 6 weeks
  the amount of air exhaled in the first second divided by all of the air exhaled during a maximal exhalation.
shortness of breath measured through borge scale of dyspnea | Changes will be assessed at baseline, 3rd week and 6th weeks measured
  shortness of breath. Changes will be assessed at baseline, 3rd week and 6th weeks measured
SGRQ questionnaire | Changes will be assessed at baseline, 3rd week and 6th weeks measured
  how breathing problems effects quality of life . Changes will be assessed at baseline, 3rd week and 6th weeks measured

CONTACTS AND LOCATIONS:
Overall Officials: Wajeeha Zia, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Mayo hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang G, Hallberg J, Um Bergstrom P, Janson C, Pershagen G, Gruzieva O, van Hage M, Georgelis A, Bergstrom A, Kull I, Linden A, Melen E. Assessment of chronic bronchitis and risk factors in young adults: results from BAMSE. Eur Respir J. 2021 Mar 4;57(3):2002120. doi: 10.1183/13993003.02120-2020. Print 2021 Mar. PMID 33184115
- [Background] Andelid K, Ost K, Andersson A, Mohamed E, Jevnikar Z, Vanfleteren LEGW, Goransson M. Lung macrophages drive mucus production and steroid-resistant inflammation in chronic bronchitis. Respir Res. 2021 Jun 7;22(1):172. doi: 10.1186/s12931-021-01762-4. PMID 34098956
- [Background] Samaha E, Vierlinger K, Weinhappel W, Godnic-Cvar J, Nohammer C, Koczan D, Thiesen HJ, Yanai H, Fraifeld VE, Ziesche R. Expression Profiling Suggests Loss of Surface Integrity and Failure of Regenerative Repair as Major Driving Forces for Chronic Obstructive Pulmonary Disease Progression. Am J Respir Cell Mol Biol. 2021 Apr;64(4):441-452. doi: 10.1165/rcmb.2020-0270OC. PMID 33524306
- [Background] Belman MJ, Thomas SG, Lewis MI. Resistive breathing training in patients with chronic obstructive pulmonary disease. Chest. 1986 Nov;90(5):662-9. doi: 10.1378/chest.90.5.662. PMID 3769566
- [Background] Kim HK, Alhammouri MT, Mokhtar YM, Pinsky MR. Estimating left ventricular contractility using inspiratory-hold maneuvers. Intensive Care Med. 2007 Jan;33(1):181-9. doi: 10.1007/s00134-006-0443-8. Epub 2006 Nov 14. PMID 17103142